CLINICAL TRIAL: NCT02759133
Title: Preoperative Localization of Infraclinical Breast Tumors: Isotopic Localization by iodine125 Seed Versus Standard Localization Using a Metal Wire: A Randomized Prospective Trial
Brief Title: Preoperative Localization of Infraclinical Breast Tumors: Isotopic Localization by iodine125 Seed Versus Standard Localization Using a Metal Wire
Acronym: IodineBreast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015/18
Record Dates: First submitted 2016-04-19; First posted 2016-05-03 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - A standard Localization technique (Active Comparator): A standard Localization technique : Metal wire as localization technique for breast cancer surgery
  Interventions: Device: Metal wire
- B - Experimental Localization technique (Experimental): Experimental Localization technique: Radioactive Iodine seed as localization technique for breast cancer surgery
  Interventions: Device: Radioactive Iodine Seed

INTERVENTIONS:
Device: Metal wire — Localization technique for breast surgery using metal wire
  Other Names: standard Localization technique
  Arms: A - A standard Localization technique
Device: Radioactive Iodine Seed — Localization technique for breast surgery using Radioactive Iodine Seed
  Other Names: Experimental Localization technique
  Arms: B - Experimental Localization technique

SUMMARY:
This is a monocentric, non-inferiority, randomized cohort study with an open 1:1 ratio comparing the impact of iodine seed tumor localization (arm B) vs. standard localization using a metal guide (arm A) on the quality of the surgical resection margins in parallel groups with an interim analysis in patients with breast cancer.

Randomization will be performed using histologic status stratification: in situ ductal /invasive lobular +/- an in situ component / invasive ductal +/- an in situ component.

DETAILED DESCRIPTION:
The widespread development of organized breast cancer screening has enabled diagnosis of nonpalpable, small-size cancer lesions (infraclinical stage). When conservative breast surgery is scheduled (tumorectomy or zonectomy), preoperative localization of the lesion is mandatory. To date, wire localization of non-palpable lesions is the most frequently used technique worldwide.

Nevertheless, this technique presents a number of drawbacks:

* it is very uncomfortable for the patient. The wire is implanted transcutaneously, crosses the skin to reach the lesion and then protrudes outside the breast, thus limiting the patient's mobility and giving rise to discomfort and even pain during movement.
* furthermore, and for the same above-mention reasons, there is a risk of the wire becoming dislodged, breaking or being disinserted during patient movements (transfer between units, pre-op shower, installation in the operating room), thus jeopardizing the quality of the planned surgery by increasing the risk of unhealthy resection margins or even of non-removal of the tumor. Cases have even been reported of intrapulmonary wire migration.
* in order to lessen these risks, the wire must be placed as late as possible before transfer to the surgical wing (the previous day at the earliest). Consequently, organizing the patient's transfer, particularly in the event of outpatient surgery (less than 12h at the hospital) becomes complicated and requires coordination between the different units in charge of preoperative management (radiology, nuclear medicine, admittance, and operating room) and early inclusion of these patients in the operating room schedule or postponement of surgery in the event of migration or displacement of the wire. These various constraints can result in a reduction of the number of patients able to benefit from outpatient management, as demonstrated by Dravet et al. Several alternative techniques have been put forward in order to overcome these difficulties, including radioguided seed localization (RSL), which consists in implanting a sealed source of radioactive iodine125 (iodine seed) inside the tumor to provide a preoperative marker which can be monitored by the surgeon using a gamma probe. The RSL technique is currently used in Europe (Netherlands), Canada and the USA.

This technique appears to offer several advantages:

* It is a simple radiologic technique performed under ultrasound or stereotaxic control, allowing accurate localization of the lesion with no risk of the marker moving or being displaced,
* It requires no special training for surgeons already skilled in the use of gamma probes in the sentinel node technique,
* It allows concomitant, interference-free performance of sentinel node surgery by means of a gamma probe able to detect specifically Tc99m and/or Iodine 125,
* It is free of organizational localization constraints limiting access to outpatient surgery, which ranks as a high priority for our governing bodies (50% of all surgeries will be performed on an outpatient basis by 2016). As the half-life of iodine seeds is 60 days, it should be possible, in theory, to insert them several days, or even several months, before surgery. In this way, patient transfer is simplified and the turnover of the operating block for outpatient management can be increased. Moreover, this localization method could also be used for tumorectomies following neoadjuvant chemotherapy,
* It presents none of the drawbacks related to patient mobility. Patient comfort is enhanced and the patient is able to move freely, with fewer risks of displacement or disinsertion, and less pain, etc.
* Patient satisfaction is higher among those women who have undergone iodine seed localization as opposed to the conventional localization techniques

Furthermore, various studies have demonstrated the safety of this technique in terms of radiation protection as radiation is minimal to the patient (equivalent to the amount received from two mammography views) as well as to the staff. Its reliability regarding the surgical excision procedure (positive or inadequate margin rates, revision surgery rates) has been demonstrated in 3 randomized studies with a high level of evidence.

Thus, in 2001, Gray et al. published the first randomized study comparing the RSL technique with the conventional wire method and showed the superiority of iodine seed localization in terms of positive margin and surgical revision rates (RSL 26% vs WL 26%, p=0.02) with no concomitant increase in tumorectomy specimen volumes or marker migration rates. More recently, Lovrics et al. (2011) and Bloomquist et al (2015) published randomized non-inferiority studies highlighting the equivalent results between these two techniques regarding the quality of tumor excision (positive margins rates in: RSL 15.1% vs WL 19% p=0.389, and in: RSL 19.4% vs 15.3%, p=0.53). In addition, the RSL method showed a significant advantage regarding operating times and pain experienced by patients during the localization procedure.

No French team has investigated this localization method on account of legal constraints. Nonetheless, it would appear that the wire localization technique does not satisfy surgical teams since another pre-operative localization technique involving injection of Tc99m into contact with the tumor has been developed over the past few years to replace the wire method. This procedure has met with little success, and has been gradually abandoned. Unfortunately, injecting Tc99m around the tumor renders the surgical procedure less precise or necessitates resecting a large segment of the gland with potentially damaging esthetic repercussions. Implantation of a sealed radioactive source such as an iodine seed helps mitigate this drawback.

This study project aims to evaluate the feasibility and safety of using 1 grain of iodine for localization purposes by means of a randomized comparative study comparing wire localization with iodine seed localization in patients presenting an in situ, biopsy-proven, non-palpable invasive or ductal breast carcinoma requiring conservative surgical management associated, or not, with an axillary procedure (SN removal or axillary curettage).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over
* Patients suffering from unifocal or in situ invasive or ductal breast cancer proven by anatomopathologic analysis (biopsy).
* Non-palpable tumor measuring at least 5 mm (minimum size deemed sufficient for the lesion to be visible by ultrasound) and ≤ 30 mm, visible by ultrasound and constituting a mass.
* Patients needing conservative first surgery management by preoperative tumor localization. For women of childbearing age, an effective contraceptive is mandatory throughout the study and up to 6 months post-operatively.
* Patients who have been made aware of the information sheet and have given their written signed informed consent.
* Patients benefitting from social health insurance coverage.

Exclusion Criteria:

* Patients with a history of homolateral breast cancer.
* Patients who have undergone neoadjuvant chemotherapy.
* Multifocal or multicentric cancer.
* Metastatic breast cancer.
* Cancer presenting in the form of microcalcifications with no visible mass.
* Vulnerable patients: pregnant or breastfeeding women, women deprived of their freedom by administrative or judicial decree, adults subject to a legal protection order or unable to give their consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2016-06; Primary Completion 2022-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
comparison of the rates of incomplete resection of the tumorectomy specimen defined according to the recommendations of the American Society of Breast Surgeons | up to 24 months

SECONDARY OUTCOMES:
surgical revision rate | up to 24 months
  Surgical revision rates are assessed by the number of surgical procedures performed for insufficient margins using the two techniques bearing in mind the analysis of systematic recuts and the surgical potential for performing revisions.
Visual Analog Score for pain | up to 24 months
Duration of surgical procedures | up to 24 months
  The duration of the localization procedure (in minutes) will be calculated from the moment the patient enters the radiology room for localization until the date of entry into the operating room. If this duration were to be extensive (several days), different groupings will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel BARRANGER, phd, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine LACASSAGNE, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barranger E, Najib B, Dejean C, Jacquinot F, Chateau Y, Chamming's F, Weitbruch D, Gosset M, Delpech Y, Gal J. Iodine125 grain isotope detection compared to standard metal guide detection for breast cancers: The IODINE BREAST, a randomised, non-inferiority trial. Eur J Surg Oncol. 2025 Dec 29;52(2):111376. doi: 10.1016/j.ejso.2025.111376. Online ahead of print. PMID 41477927
- See also: Related Info — http://www.centreantoinelacassagne.org/